CLINICAL TRIAL: NCT01775774
Title: A Phase 1 Multi-center Clinical Trial of Allogeneic Bone Marrow-derived Human Mesenchymal Stem Cells for the Treatment of Acute Respiratory Distress Syndrome
Brief Title: Human Mesenchymal Stem Cells For Acute Respiratory Distress Syndrome
Acronym: START
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Michael A. Matthay (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Massachusetts General Hospital (Other); Stanford University (Other); University of Pittsburgh (Other); University of Minnesota (Other)
Responsible Party: Sponsor-Investigator, Michael A. Matthay, Prinicpal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARDS MSC 001; 1U01HL108713-01 (NIH)
Record Dates: First submitted 2013-01-18; First posted 2013-01-25 (Estimated); Results first posted 2017-08-14 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-05

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Acute Respiratory Distress Syndrome; Acute Lung Injury; Allogeneic Bone Marrow-Derived Human Mesenchymal Stem Cells
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Allogeneic Bone Marrow-Derived Human Mesenchymal Stem Cells (Experimental): A dose-escalation with 3 cohorts with 3 subjects/cohort who receive doses of 1, 5 and 10 million cells/kg predicted body weight (PBW). Proceed from lower dose to next higher dose if no safety concerns for each cohort.
  Interventions: Biological: Allogeneic Bone Marrow-Derived Human Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Allogeneic Bone Marrow-Derived Human Mesenchymal Stem Cells — Allogeneic Bone Marrow-Derived Human Mesenchymal Stem Cells will be administered intravenously.

SUMMARY:
This is a Phase 1, open label, dose escalation, multi-center clinical trial of Allogeneic Bone Marrow-Derived Human Mesenchymal Stem Cells (hMSCs) for the treatment of Acute Respiratory Distress Syndrome (ARDS). The purpose of this study is to assess the safety of hMSCs in patients with ARDS.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the safety of intravenous infusion of Allogeneic Bone Marrow-Derived Human Mesenchymal Stem Cells (hMSCs) in patients with ARDS.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for inclusion if they meet all of the below criteria. Criteria 1-3 must all be present within a 24-hour time period and at the time of enrollment:

Acute onset (defined below) of:

1. A need for positive pressure ventilation by an endotracheal or tracheal tube with a PaO2/FiO2 ratio < 200 with at least 8 cm H2O positive end-expiratory airway pressure (PEEP)
2. Bilateral infiltrates consistent with pulmonary edema on frontal chest radiograph
3. No clinical evidence of left atrial hypertension for bilateral pulmonary infiltrates.

In addition to meeting inclusion criteria, enrollment must occur within 96-hours of first meeting ARDS criteria per the Berlin definition of ARDS.

Exclusion Criteria:

1. Age less than 18 years
2. Greater than 96 hours since first meeting ARDS criteria per the Berlin definition of ARDS
3. Pregnant or breast-feeding
4. Prisoner
5. Presence of any active malignancy (other than non-melanoma skin cancer) that required treatment within the last 2 years
6. Any other irreversible disease or condition for which 6-month mortality is estimated to be greater than 50%
7. Moderate to severe liver failure (Childs-Pugh Score > 12)
8. Severe chronic respiratory disease with a PaCO2 > 50 mm Hg or the use of home oxygen
9. Patient, surrogate, or physician not committed to full support (exception: a patient will not be excluded if he/she would receive all supportive care except for attempts at resuscitation from cardiac arrest).
10. Major trauma in the prior 5 days
11. Lung transplant patient
12. No consent/inability to obtain consent
13. Moribund patient not expected to survive 24 hours
14. WHO Class III or IV pulmonary hypertension
15. Documented deep venous thrombosis or pulmonary embolism within past 3 months
16. No arterial line/no intent to place an arterial line
17. No intent/unwillingness to follow lung protective ventilation strategy or fluid management protocol
18. Currently receiving extracorporeal life support (ECLS) or high-frequency oscillatory ventilation (HFOV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-07; Primary Completion 2014-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of California San Francisco Medical Center, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wilson JG, Liu KD, Zhuo H, Caballero L, McMillan M, Fang X, Cosgrove K, Vojnik R, Calfee CS, Lee JW, Rogers AJ, Levitt J, Wiener-Kronish J, Bajwa EK, Leavitt A, McKenna D, Thompson BT, Matthay MA. Mesenchymal stem (stromal) cells for treatment of ARDS: a phase 1 clinical trial. Lancet Respir Med. 2015 Jan;3(1):24-32. doi: 10.1016/S2213-2600(14)70291-7. Epub 2014 Dec 17. PMID 25529339
- [Derived] Liu KD, Wilson JG, Zhuo H, Caballero L, McMillan ML, Fang X, Cosgrove K, Calfee CS, Lee JW, Kangelaris KN, Gotts JE, Rogers AJ, Levitt JE, Wiener-Kronish JP, Delucchi KL, Leavitt AD, McKenna DH, Thompson BT, Matthay MA. Design and implementation of the START (STem cells for ARDS Treatment) trial, a phase 1/2 trial of human mesenchymal stem/stromal cells for the treatment of moderate-severe acute respiratory distress syndrome. Ann Intensive Care. 2014 Jul 3;4:22. doi: 10.1186/s13613-014-0022-z. eCollection 2014. PMID 25593740
- [Derived] Asmussen S, Ito H, Traber DL, Lee JW, Cox RA, Hawkins HK, McAuley DF, McKenna DH, Traber LD, Zhuo H, Wilson J, Herndon DN, Prough DS, Liu KD, Matthay MA, Enkhbaatar P. Human mesenchymal stem cells reduce the severity of acute lung injury in a sheep model of bacterial pneumonia. Thorax. 2014 Sep;69(9):819-25. doi: 10.1136/thoraxjnl-2013-204980. Epub 2014 Jun 2. PMID 24891325

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This dose-escalation Phase 1 clinical trial with 3 cohorts with 3 subjects/cohort was performed in 7 centers in USA between July 2013 to January 2014.
Groups:
- Human Mesenchymal Stem Cells 1 Million Cells/kg PBW; Human Mesenchymal Stem Cells 5 Million Cells/kg PBW; Human Mesenchymal Stem Cells 10 Million Cells/kg PBW: Allogeneic Bone Marrow-Derived Human Mesenchymal Stem Cells were administered intravenously into the 3 planned dosing cohorts.
Period: Overall Study
Arm/Group | Human Mesenchymal Stem Cells 1 Million Cells/kg PBW | Human Mesenchymal Stem Cells 5 Million Cells/kg PBW | Human Mesenchymal Stem Cells 10 Million Cells/kg PBW
Started | 3 | 3 | 3
Completed | 3 | 3 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Mesenchymal Stem Cells 5 Million Cells/kg PBW; Mesenchymal Stem Cells 10 Million Cells/kg PBW: Allogeneic Bone Marrow-Derived Human Mesenchymal Stem Cells were administered intravenously into the 3 planned dosing cohorts.
- Total: Total of all reporting groups
Arm/Group | Human Mesenchymal Stem Cells 1 Million Cells/kg PBW | Mesenchymal Stem Cells 5 Million Cells/kg PBW | Mesenchymal Stem Cells 10 Million Cells/kg PBW | Total
Number analyzed (Participants) | 3 | 3 | 3 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 3 | 7
  >=65 years | 1 | 1 | 0 | 2
Age, Continuous [Mean (Full Range); unit: years] | 58.0 [29 to 86] | 58.3 [46 to 67] | 48.3 [38 to 55] | 54.9 [29 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 1 | 7
  Male | 0 | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 3 | 1 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 3 | 2 | 7
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 9
APACHE III Score [Mean (Full Range); unit: scores on a scale] — Acute Physiology and Chronic Health Evaluation III score, a severity-of-disease classification system. Higher score predicts worse clinical outcome. The scale of APACHE III is 0 - 299, where 0 = best outcome and 299 = worst outcome.
  scores on a scale | 91.7 [62 to 111] | 89.7 [64 to 115] | 88.3 [54 to 108] | 89.9 [54 to 115]
Primary cause of ARDS [Number; unit: participants]
  Pneumonia | 1 | 1 | 2 | 4
  Aspiration | 1 | 2 | 0 | 3
  Sepsis | 0 | 0 | 1 | 1
  Pre-eclampsia | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Pre-specified Infusion Associated Adverse Events
Description: Any of the following occurring within 6 h of mesenchymal stem-cell infusion:
  * Addition of a third vasopressor or an increase in vasopressor dose greater than or equal to the following:
  * Norepinephrine: 10 μg per min
  * Phenylephrine: 100 μg per min
  * Dopamine: 10 μg/kg per min
  * Epinephrine: 0·1 μg/kg per min
  * Hypoxaemia requiring an increase in the fraction of inspired oxygen of ≥0·2 and increase in positive end-expiratory airway pressure level of 5 cm H2O or more to maintain transcutaneous oxygen saturations in the target range of 88-95%
  * New cardiac arrhythmia requiring cardioversion
  * New ventricular tachycardia, ventricular fi brillation, or asystole
  * A clinical scenario consistent with transfusion incompatibility or transfusion-related infection
  * Cardiac arrest or death within 24 h of mesenchymal stem-cell infusion
Time Frame: 24 hours
Measure: Number; unit: participants
Groups:
- Human Mesenchymal Stem Cells: 1 Million Cellls/kg PBW; Human Mesenchymal Stem Cells: 5 Million Cellls/kg PBW; Human Mesenchymal Stem Cells: 10 Million Cellls/kg PBW: Allogeneic Bone Marrow-Derived Human Mesenchymal Stem Cells were administered intravenously into the 3 planned dosing cohorts.
Arm/Group | Human Mesenchymal Stem Cells: 1 Million Cellls/kg PBW | Human Mesenchymal Stem Cells: 5 Million Cellls/kg PBW | Human Mesenchymal Stem Cells: 10 Million Cellls/kg PBW
Number analyzed (Participants) | 3 | 3 | 3
participants | 0 | 0 | 0

2. Secondary Outcome: Incidence of Severe Adverse Events (SAEs)
Description: The number of participants with a severe adverse event during the study was assessed.
Time Frame: Investigators conducted daily assessments for the presence of adverse events (AE) from enrollment through study day 28 or hospital discharge, whichever occurred first.
Measure: Number; unit: participants
Arm/Group | Human Mesenchymal Stem Cells: 1 Million Cellls/kg PBW | Human Mesenchymal Stem Cells: 5 Million Cellls/kg PBW | Human Mesenchymal Stem Cells: 10 Million Cellls/kg PBW
Number analyzed (Participants) | 3 | 3 | 3
participants | 2 | 1 | 0

3. Secondary Outcome: Ventilator Free Days at Study Day 28
Description: Ventilator Free Days (VFDs) to day 28 were defined as the number of days from the time of initiating unassisted breathing to day 28 after randomization, assuming survival for at least two consecutive calendar days after initiating unassisted breathing and continued unassisted breathing to day 28. If a subject received assisted breathing at day 27 or died prior to day 28, a value of zero VFDs was given.
Time Frame: time of initiating unassisted breathing to day 28
Measure: Median (Full Range); unit: day
Arm/Group | Human Mesenchymal Stem Cells: 1 Million Cellls/kg PBW | Human Mesenchymal Stem Cells: 5 Million Cellls/kg PBW | Human Mesenchymal Stem Cells: 10 Million Cellls/kg PBW
Number analyzed (Participants) | 3 | 3 | 3
day | 18 [0 to 24] | 22 [0 to 27] | 20 [12 to 26]

4. Secondary Outcome: Duration of Vasopressor Use (Days)
Description: Days on vasopressor to day 28 after study enrollment
Time Frame: 28 days
Measure: Median (Full Range); unit: day
Arm/Group | Human Mesenchymal Stem Cells: 1 Million Cellls/kg PBW | Human Mesenchymal Stem Cells: 5 Million Cellls/kg PBW | Human Mesenchymal Stem Cells: 10 Million Cellls/kg PBW
Number analyzed (Participants) | 3 | 3 | 3
day | 4 [0 to 10] | 2 [0 to 3] | 0 [0 to 0]

5. Secondary Outcome: ICU Free Days to Day 28
Time Frame: 28 days after study enrollment
Measure: Median (Full Range); unit: day
Arm/Group | Human Mesenchymal Stem Cells: 1 Million Cellls/kg PBW | Human Mesenchymal Stem Cells: 5 Million Cellls/kg PBW | Human Mesenchymal Stem Cells: 10 Million Cellls/kg PBW
Number analyzed (Participants) | 3 | 3 | 3
day | 14 [0 to 24] | 21 [0 to 26] | 18 [9 to 22]

6. Secondary Outcome: Hospital Survival to Day 60
Description: The number of subjects alive at study day 60. Those subjects discharged home prior to day 60 were counted as alive at day 60.
Time Frame: 60 days after randomization
Measure: Number; unit: participants
Arm/Group | Human Mesenchymal Stem Cells: 1 Million Cellls/kg PBW | Human Mesenchymal Stem Cells: 5 Million Cellls/kg PBW | Human Mesenchymal Stem Cells: 10 Million Cellls/kg PBW
Number analyzed (Participants) | 3 | 3 | 3
participants | 2 | 2 | 3

7. Secondary Outcome: Mortality at Hospital Discharge
Description: The number of patients expired at hospital discharge.
Time Frame: From study enrollment to Hospital discharge
Measure: Number; unit: participants
Arm/Group | Human Mesenchymal Stem Cells: 1 Million Cellls/kg PBW | Human Mesenchymal Stem Cells: 5 Million Cellls/kg PBW | Human Mesenchymal Stem Cells: 10 Million Cellls/kg PBW
Number analyzed (Participants) | 3 | 3 | 3
participants | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Human Mesenchymal Stem Cells: 1 Million Cells/kg PBW; Human Mesenchymal Stem Cells: 5 Million Cells/kg PBW; Human Mesenchymal Stem Cells: 10 Million Cells/kg PBW: Allogeneic Bone Marrow-Derived Human Mesenchymal Stem Cells will be administered intravenously.
Arm/Group | Human Mesenchymal Stem Cells: 1 Million Cells/kg PBW | Human Mesenchymal Stem Cells: 5 Million Cells/kg PBW | Human Mesenchymal Stem Cells: 10 Million Cells/kg PBW
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Human Mesenchymal Stem Cells: 1 Million Cells/kg PBW (N=3) | Human Mesenchymal Stem Cells: 5 Million Cells/kg PBW (N=3) | Human Mesenchymal Stem Cells: 10 Million Cells/kg PBW (N=3)
Multiorgan failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Infarcts of kidneys, spleen and brain (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Human Mesenchymal Stem Cells: 1 Million Cells/kg PBW (N=3) | Human Mesenchymal Stem Cells: 5 Million Cells/kg PBW (N=3) | Human Mesenchymal Stem Cells: 10 Million Cells/kg PBW (N=3)
Elevated liver function tests (Hepatobiliary disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No